CLINICAL TRIAL: NCT05065047
Title: Belantamab Mafadotin Maintenance Therapy After Salvage Autologous Hematopoietic Cell Transplantation in Patients With Relapse Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1059; NCI-2021-09412 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-08-25; First posted 2021-10-01 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belantamab mafodotin (Experimental): belantamab mafodotin by vein over 30 minutes every 8 weeks
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Belantamab mafodotin — Given by IV

SUMMARY:
The goal of this clinical research study is to learn if belantamab mafodotin (Blenrep) can help to prevent multiple myeloma (MM) from coming back after patients have had an autologous stem cell transplant (AutoSCT). The safety of this drug after transplant will also be studied

DETAILED DESCRIPTION:
Primary Objective:

To determine the safety and tolerability of belantamab maintenance therapy after auto-HCT.

Secondary Objectives:

* To estimate the complete remission rate (CRR) as defined by the International Myeloma Working Group (IMWG) criteria (Appendix A.) within 9 months post salvage autotransplant with single agent belantamab mafodotin maintenance therapy starting approximately 3 months post salvage auto-transplant in patients with relapsed myeloma.
* To evaluate progression-free survival (PFS) and overall survival (OS) (from the data of initiation of maintenance therapy assessed up to 2 years)
* To discover the impact of belantamab mafodotin on graft function and immune reconstitution.
* • To assess minimal residual disease status (FDA approved MRD assay by flow cytometry - MRD measured down to 1 in 1 million cells, <106) after at 6 months and 1, 2, and 3 years after initiation of maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory multiple myeloma. Eligible patients will be enrolled in the protocol no less than 60 days and must be initiated no longer than 180 days (± 2 weeks) post ASCT. Patient's transplant may be either transplantation naïve or with a history of previous autologous transplant.
2. Patients who have had two or more lines of therapy consisting of at least one of three agents including a proteasome inhibitor or an immunomodulatory agent or an anti-CD38 targeting therapy.

   Note:

   a) Induction therapy, autologous stem cell transplantation (ASCT) & maintenance therapy if given sequentially without intervening progressive disease (PD) are considered one line of therapy. b) Refractory MM may be defined as disease that is refractory to treatment while on therapy or that shows progression within 60 days of the last therapy.
3. Disease status, partial response, or better.
4. Age ≥ 18-year and ≤ 75-year. English and non-English speaking patients are eligible.
5. Platelet count ≥ 50,000/mm3 & Hemoglobin ≥ 8 g/dL, ANC ≥ 1.0 × 109/L
6. Karnofsky Performance Status (KPS) >70 (Appendix B.).
7. Adequate organ function (ALT ≤ 2.5 ULN; Total bilirubin ≤ 1.5 ULN or total bilirubin

   * 1.5 ULN with direct bilirubin ≤ 35%; estimated glomerular filtration rate ≥30 mL/min per 1.73 m2
8. Participants must not be pregnant or lactating
9. Female participants: contraceptive use should be consistent with institutional guidelines regarding the methods of contraception for those participating in clinical studies.

A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

1. Is not a woman of childbearing potential (WOCBP) OR
2. Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency (as described in Appendix C.), during the intervention period and for at least 4 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relation to the first dose of the study intervention.

   A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 72 hours before the first dose of the study intervention.

   Nonchildbearing potential is defined as follows (by other than medical reasons):

   • ≥45 years of age and has not had menses for >1 year

   • Patients who have been amenorrhoeic for <2 years without a history of a hysterectomy and oophorectomy must have a follicle-stimulating hormone value in the postmenopausal range upon screening evaluation

   • Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. 10. Male participants: contraceptive use should be consistent with institutional guidelines regarding the methods of contraception for those participating in clinical studies.

   Male participants are eligible to participate if they agree to the following during the intervention period and for 6 months after the last dose of study treatment to allow for clearance of any altered sperm:
   * Refrain from donating sperm

   PLUS either:
   * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent.

   OR

   • Must agree to use contraception/barrier as detailed below: Agree to use a male condom, even if they have undergone a successful vasectomy and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as to when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.

   Exclusion Criteria:

   1. Current corneal epithelial disease (except mild punctate keratopathy). 2. Participant must not use contact lenses while participating in this study. 3. Ongoing Grade 2 or higher peripheral neuropathy or neuropathic pain. 4. Participants who are using an investigational drug or approved systemic anti-myeloma therapy (including systemic steroids) within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug.

   5. Participants who have current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia (serum albumin < 3.0 gm/dl), esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria 6. Participants who have presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfil inclusion criteria 7. Participants who have received prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drugs.

   8. Participants who have had major surgery ≤ 4 weeks before initiating study treatment.

   9. Participants who have any evidence of active mucosal or internal bleeding. 10. Participants who have known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.

   11. Participants who have an active infection requiring treatment 12. Participants who have evidence of cardiovascular risk, including any of the following:

a) Evidence of current clinically significant uncontrolled and/or untreated arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block.

b) History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within three (3) months of screening.

c) Class III or IV heart failure as defined by the New York Heart Association functional classification system.

d) Uncontrolled hypertension. 13. Participants who have known HIV infection, unless the participant can meet all of the following criteria:

* Established anti-retroviral therapy (ART) for at least 4 weeks and HIV viral load <400 copies/mL
* CD4+ T-cell (CD4+) counts ≥350 cells/uL
* No history of AIDS-defining opportunistic infections within the last 12 months 14. Participant must not have presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb) at screening or within 3 months prior to first dose of study treatment. Note: presence of Hep B surface antibody (HBsAb) indicating previous vaccination will not exclude a participant.

  15. Participant must not have positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment.

Note: Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained.

Note: Hepatitis RNA testing is optional and participants with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing.

16. Participant must not have invasive malignancies other than disease under study, unless the second malignancy has been medically stable for at least 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Participants with curatively treated non-melanoma skin cancer may be enrolled without a 2-year restriction.

17. Prior allogeneic stem cell transplant. NOTE: Participants who have undergone syngeneic transplant will be allowed only if no history of or no currently active GvHD.

18. Symptomatic amyloidosis, active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasmaproliferative disorder, skin changes) or active plasma cell leukaemia at the time of screening.

19. Patients with cognitive impairments and/or any serious unstable pre-existing medical condition or psychiatric disorder that can interfere with safety or with obtaining informed consent or compliance with study procedures. Informed Consent Process. The informed consent process will begin at recognition of subject eligibility, and consent will be obtained per Institutional practices before study therapy is initiated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0, Change From Baseline in Pain Scores on the Visual Analog Scale at 6 Weeks | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Saini, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT05065047/ICF_000.pdf